CLINICAL TRIAL: NCT01283672
Title: Acute Heart Health Benefits of Whole Grain Barley and Oats in Healthy Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Kellogg Company (Industry)
Responsible Party: David J. Baer, USDA
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS33
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Cardiovascular Disease
Keywords: Whole grains; Barley; Oats; Cardiovascular disease; Postprandial lipid metabolism; Endothelial function; Risk of cardiovascular disease in healthy men and women
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Controlled diet with whole grain barley, whole grain oats, or low grain diet — Participants will consume a standardized diet for 3 days prior to the treatment intervention meal. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet. Participants will be instructed to eat all foods and only foods provided to them, with the exception of water, coffee, tea, and diet soda.

SUMMARY:
The objectives of this study are the following: 1) to determine the acute effect of whole grain barley on risk factors of cardiovascular disease compared to a diet low in whole grain, and 2) to compare the effects of whole grain barley to those of whole grain oats to determine if the response to these two grains is similar.

DETAILED DESCRIPTION:
Whole grains contain bioactive components that may contribute to reduced risk of cardiovascular disease, and there may be significant differences among whole grain sources with respect to ability to alter biomarkers of cardiovascular disease. This acute study is designed to determine if whole grain barley improves postprandial lipid metabolism and improves endothelial function. Further, we will determine if acute consumption of whole grain barley versus acute consumption of whole grain oats results in differential response with respect to biomarkers of cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 25-70 years
* Body mass index (BMI) ≥ 19 and ≤ 38
* Willingness and ability to make scheduled appointments at clinical site as required by study protocol

Exclusion Criteria:

* Do not regularly consume breakfast or dislike cereal for breakfast
* Known (self-reported) allergy or adverse reaction to grains (e.g., wheat, gluten, barley)
* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides > 300 mg/dL
* Fasting glucose > 126 mg/dL
* Use of cholesterol lowering medication
* Blood pressure > 180/100 or hypertension treated with calcium channel blockers, direct acting vasodilators, or beta blockers
* Fingernails longer than 0.25 inch beyond the finger tip, or unwillingness to cut fingernails to this length during endothelial function testing
* History of bariatric or certain other surgeries related to weight control
* History of major surgery within 3 months of enrollment
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 months prior to the intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 6 months
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Lipid Tolerance Test | After 3 consecutive days of controlled feeding.
  Participants will come in after a 12-hour fast for a lipid tolerance test. Specifically, participants will consume a treatment breakfast meal and blood samples will be collected 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 360, and 420 minutes following ingestion of the treatment meal.
EndoPAT | After 3 consecutive days of controlled feeding
  Endothelial function will be assessed by measuring endothelium-dependent flow mediated dilation of the peripheral bed (EndoPAT, Itamar Medical, Israel). Immediately after the test, a blood sample will be collected for measurement of serum triglycerides.

SECONDARY OUTCOMES:
Genetic testing | After 3 consecutive days of controlled feeding
  Blood will be used to test for genetic traits that may influence nutrient metabolism and also traits reflecting the mechanisms that may be influenced by the intervention.
Microarray and targeted gene expression testing | After 3 consecutive days of controlled feeding
  Blood samples will be used to test how the intervention affects gene expression. Global gene expression will be performed for a complete survey of the RNA response to the intervention, and targeted gene expression will be performed to confirm the findings of the global gene expression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David J Baer, PhD, Principal Investigator — US Department of Agriculture
Locations (1):
- US Department of Agriculture Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States